CLINICAL TRIAL: NCT06419595
Title: Screening and Support for Youth
Brief Title: Screening and Support for Youth (SASY)
Acronym: SASY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge Health Alliance (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Exploratory 1; PAR-24-210 (Other Grant/Funding Number: NIMH)
Record Dates: First submitted 2024-05-14; First posted 2024-05-17 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Adolescent Health; Minority Health; Mental Health; Community Health Services
MeSH Terms: conditions — Psychological Well-Being | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Recruitment by Research Coordinator (RC) (Other): Study participants will be randomized for recruitment follow up by research team RC.
  Interventions: Behavioral: Behavioral: Screening and Support for Youth (SASY) Multi-component Platform: includes screening, feedback, single session intervention, and resource information
- Recruitment by EYE (Other): Study participants will be randomized for recruitment follow up by the EYE peer group (community youth research group)
  Interventions: Behavioral: Behavioral: Screening and Support for Youth (SASY) Multi-component Platform: includes screening, feedback, single session intervention, and resource information

INTERVENTIONS:
Behavioral: Behavioral: Screening and Support for Youth (SASY) Multi-component Platform: includes screening, feedback, single session intervention, and resource information — Description: Description: Participants who interact with a QR code and express interest in participating will be randomized to receive either: 1) recruitment from a Research Coordinator (standard research staff approach) or 2) recruitment from an EYE for Prevention Youth Researcher. The process of consent, screening, providing feedback, and offering access to a Single Session Intervention and information on additional resources (per scoring on the screening into Tier 1 (low risk/normal), 2 (moderate/at risk), or 3 (high/clinical risk): Tier 1 = screening+feedback; Tier 2=screening+feedback+SSI; Tier 3=screening+feedback+SSI+resource information) will be the same in each group. The randomization is simply changing who provides the process and platform to the participant.
  Arms: Recruitment by EYE
Behavioral: Behavioral: Screening and Support for Youth (SASY) Multi-component Platform: includes screening, feedback, single session intervention, and resource information — Description: Description: Participants who interact with a QR code and express interest in participating will be randomized to receive either: 1) recruitment from a Research Coordinator (standard research staff approach) or 2) recruitment from an EYE for Prevention Youth Researcher. The process of consent, screening, providing feedback, and offering access to a Single Session Intervention and information on additional resources (per scoring on the screening into Tier 1 (low risk/normal), 2 (moderate/at risk), or 3 (high/clinical risk): Tier 1 = screening+feedback; Tier 2=screening+feedback+SSI; Tier 3=screening+feedback+SSI+resource information) will be the same in each group. The randomization is simply changing who provides the process and platform to the participant.
  Arms: Recruitment by Research Coordinator (RC)

SUMMARY:
To adapt the Screening and Support for Youth (SASY) intervention and approach to recruitment for racial, ethnic and linguistic diverse youth aged 12-17 in the Denver Health catchment area

DETAILED DESCRIPTION:
To adapt the Screening and Support for Youth (SASY) intervention and approach to recruitment for racial, ethnic and linguistic diverse youth aged 12-17 in the Denver Health catchment area.

Includes the recruitment of 220 youth (170 from schools/community and 50 hard-to-reach).

170 participants will be recruited by QR codes available on flyers that will be distributed in schools and community settings. This group will then be randomized to either follow up with the Engaging Youth Expertise for Prevention (EYE) or one of the study team's Research Coordinators (RC) and either EYE or the RC will carry out the assent/consent process with youth and their parents/guardians. For the subsequent (non-randomized) group of 50 hard-to-reach participants, the EYE team will utilize various methods for recruitment, and coordinate the assent/consent process with youth and their parents/guardians.

All 200 participants will be offered a SASY screening which will include the K-CAT, Weiss Functional Impairment Scale (WFIRS-S), CAT-MH social determinants of health (SDOH), and assessment of current mental health treatment. All survey instruments will be delivered via REDCap. Each participant will be assigned a record identification (ID) and an acrostic, so their data can not be identifiable during analysis. All data will stay within the Cambridge Health Alliance (CHA) firewall and only the study team will have access to the results. These products are available in English and Spanish.

A clinical risk score is generated by an algorithm combining symptoms and functional impairment based on national norms. Tier 1 is within normal, Tier 2 is at clinical risk, and Tier 3 is clinically ill. All participants will receive a motivational feedback session to discuss the results of the screening. The discussion will focus on the participant's reflections on how they feel, their perception of their symptoms and functioning, what changes they wish to make in their life, and what might support that change. The feedback will be given to the teens using non-clinical and non-research terms based upon the students' responses on the screening measures. Tier 1 participants will be offered screening and feedback on the screening results. Tier 2 participants will be offered screening, feedback on the screening results and a single session intervention (SSI). Tier 3 participants will be offered screening, feedback on the screening results, a single session intervention and information on community resources. The SSI will be accessed by a unique link provided to the participants, and includes several modules to choose from that participants can complete on their own and at their own pace.

All participants will be invited for a follow-up survey at 1 month following initial screening. The follow-up survey will re-assess the KCAT and WFIRS, therapeutic alliance, and engagement in mental health treatment or behavioral interventions.

All participants will be offered a $20 incentive for the initial screening and $20 for completing the follow-up survey.

ELIGIBILITY:
Inclusion Criteria:

* 12 to 17 year old teens

Exclusion Criteria:

* younger than 12 or older than 17

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220 (Estimated)
Dates: Start 2026-11-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Completion of Single session intervention | 1 month following initial screening
  Number and proportion of participants in Tiers 2 and 3 that start and/or complete the single session intervention. This will be a measure of engagement in services.
Participation | Immediate at time of enrollment
  Total number and proportion of 12-17 year olds recruited by the Research Coordinator vs. EYE Youth Researchers; also will examine this by proportion racial, ethnic and linguistic (REL) minoritized youth who participate (comparing Research Coordinator vs. EYE)

SECONDARY OUTCOMES:
K-CAT/WFIRS scores - preliminary effectiveness | 1 month following initial screening
  Change on the K-CAT/WFIRS scores between time of screening (pre-) and post-intervention (SSI as the intervention) for Tiers 2 and 3
Therapeutic Alliance | 1 month following initial screening
  Measure of therapeutic alliance with a) recruitment, screening, feedback and b) SSI.
Engagement in Mental Health Treatment/Behavioral Change Activities | 1 month following initial screening
  Self-reported measure of engagement for youth who scored in Tier 3 (and were provided SSI + resources).

CONTACTS AND LOCATIONS:
Overall Officials: Laura Podewils, Principal Investigator — Denver Health and Hospital Authority

IPD SHARING:
Plan to Share IPD: No
Information will contain health insurance portability and accountability act (HIPAA) identifiers